CLINICAL TRIAL: NCT01624350
Title: MASERATI 100 - A Prospective, Multi-center, Post-mArket, Single-arm obsERvATIonal Study to Collect Clinical Outcome Data on the Use of Permacol™ Collagen Paste in the Treatment of Anorectal Fistulas
Brief Title: A Prospective, Multi-center, Observational Study of the Use of Permacol™ Collagen Paste to Treat Anorectal Fistulas
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVPERP0200
Record Dates: First submitted 2012-06-15; First posted 2012-06-20 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Anorectal Fistulas
Keywords: Anorectal Fistulas
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Permacol collagen paste — Collagen paste intended to reinforce soft tissue where filling is required such as to repair fistulas, including anal and rectal fistulas.

SUMMARY:
This will be a prospective, multi-center, post-market, single arm observational study to collect clinical outcome data on the use of Permacol™ Collagen Paste in the treatment of anorectal fistulas.

The subjects will have baseline and day of surgery visits performed, and then subjects will return to the investigator for evaluation of defect and safety related morbidities at follow up visits scheduled at 1 month, 3 months, 6 months and 12 months post-surgery.

DETAILED DESCRIPTION:
The study will enroll 100 subjects at up to 10 centers throughout the European Union. The expected duration of the enrollment period is approximately 9 months. The duration of each subject's participation in the study will be approximately one year. However, at sites where the routine follow-up period is greater than one year, subjects may be followed for up to 36 months at their surgeon's discretion if they agree to it.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects age 18 or older
2. Subjects diagnosed with a solitary tract anorectal fistula of cryptoglandular origin

Key Exclusion Criteria:

1. History or suspicion of Inflammatory Bowel Disease (i.e.Crohn's Disease, Ulcerative Colitis)
2. Subjects with secondary tracts, horseshoe fistulas, ano/recto-vaginal fistulas, or rectourethral fistulas
3. Indication of an actively infected fistula/abscess (acute sepsis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who meet the eligibility criteria that are planned to undergo surgical treatment for anorectal fistulas with Permacol™ Collagen Paste and agree to 12 months of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Giordano, MD, FRCS, Principal Investigator — Whipps Cross University Hospital
Locations (10):
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus C
- Italy (3):
  - Casa di Cura PIO X, Milan
  - AO S.Maria degli Angeli, S.S.D. Degenze Brevi 1^ 2^ Chirurgia Ginecologia e Urologia, Pordenone
  - University of Rome Tor Vergata, Surgery-Policlinico Tor Vergata, Rome
- United Kingdom (5):
  - Ninewells Hospital & Medical School, Dundee
  - Leicester General Hospital, Leicester
  - King's College Hospital, London
  - Whipps Cross University Hospital, London
  - Royal Victoria Infirmary, Newcastle

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Permacol Collagen Paste
Started | 100
Completed | 75
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Permacol Collagen Paste
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.68)
Gender [Count of Participants; unit: Participants]
  Female | 30
  Male | 70
Region of Enrollment [Number; unit: participants]
  Denmark | 15
  United Kingdom | 52
  Italy | 33

OUTCOME MEASURES:

1. Primary Outcome: Fistula Healing in Patients at 6 Months Following Surgery
Description: Clinical assessment of fistula healing as defined by 1) no discharge from the fistula and 2) the external opening has closed.
Time Frame: 6 months
Population: Number of participants analyzed includes patients who had their assessment performed and the final assessment of patients who exited from the study early.
Measure: Number; unit: percentage of participants
Arm/Group | Permacol Collagen Paste
Number analyzed (Participants) | 97
percentage of participants
  Yes | 56.7
  No | 43.3

2. Secondary Outcome: Fistula Healing in Patients at 3 and 12 Months Following Surgery
Description: as for outcome 1
Time Frame: 3 months and 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Permacol Collagen Paste - 3 Month Follow up | Permacol Collagen Paste - 12 Month Follow up
Number analyzed (Participants) | 94 | 99
percentage of patients
  Yes | 53.2 [42.6 to 63.6] | 53.5 [43.2 to 63.6]
  No | 46.8 [42.6 to 63.6] | 46.5 [43.2 to 63.6]

3. Secondary Outcome: Participant Response to Quality of Life EQ-5D Questionnaire
Description: Quality of Life by EQ-5D questionnaire is a standardized measure of health status. It is a 25-item questionnaire that measures quality of life of patients pre and post surgery in the following categories: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each category has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Time Frame: Baseline, and 3 months, 6 months and 12 months post op
Population: Number analyzed include participants who completed questionnaire.
Measure: Number; unit: participants
Arm/Group | Baseline - Pre-operatively | Permacol Collagen Paste - 3 Month Post-op | Permacol Collagen Paste - 6 Month Post-op | Permacol Collagen Paste - 12 Month Post-op
Number analyzed (Participants) | 97 | 88 | 79 | 74
participants
  I have no problems in walking about | 74 | 77 | 76 | 72
  I have slight problems in walking about | 13 | 7 | 2 | 0
  I have moderate problems in walking about | 10 | 3 | 0 | 1
  I have severe problems in walking about | 0 | 1 | 0 | 1
  I am unable to walk about | 0 | 0 | 1 | 0
  I have no problems washing or dressing myself | 87 | 84 | 78 | 72
  I have slight problems washing or dressing myself | 7 | 3 | 0 | 1
  I have moderate problems washing or dressing mysel | 1 | 1 | 1 | 1
  I have severe problems washing or dressing myself | 1 | 0 | 0 | 0
  I am unable to wash or dress myself | 1 | 0 | 0 | 0
  I have no problems doing my usual activities | 72 | 69 | 72 | 63
  I have slight problems doing my usual activities | 13 | 12 | 6 | 9
  I have moderate problems doing my usual activities | 8 | 6 | 0 | 1
  I have severe problems doing my usual activities | 4 | 1 | 1 | 1
  I have no pain or discomfort | 38 | 46 | 52 | 49
  I have slight pain or discomfort | 44 | 31 | 22 | 20
  I have moderate pain or discomfort | 13 | 10 | 4 | 3
  I have severe pain or discomfort | 2 | 1 | 0 | 1
  I have extreme pain or discomfort | 0 | 0 | 1 | 1
  I am not anxious or depressed | 63 | 69 | 67 | 56
  I am slightly anxious or depressed | 24 | 13 | 9 | 13
  I am moderately anxious or depressed | 8 | 6 | 2 | 4
  I am severely anxious or depressed | 1 | 0 | 0 | 0
  I am extremely anxious or depressed | 1 | 0 | 1 | 1

4. Secondary Outcome: Fecal Incontinence
Description: Fecal Incontinence change from baseline as measured by CCF-FI questionnaire. This questionnaire is a summed score of 5 individual parameters (frequency of incontinence to gas, liquid solid, of need to wear pad, and of lifestyle changes) It is measured from a patient-completed questionnaire with each parameter given a score from 0 to 4, with 0 indicating its absence and 4 indicating daily presence. These values are added to give a total score ranging from 0 to 20 (0 indicating perfect control, 10-15 indicating moderate incontinence, and greater than 15 indicating severe incontinence.
Time Frame: 3 months, 6 months and 12 months
Population: The CCF-FI score was calculated if a score was ticked for each of the five types of incontinence. If a patient had a type of incontinence with a missing score, then the CCF-FI score was not calculated. Change = Value and Month X - Value at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Permacol Collagen Paste - 3 Month Post-op | Permacol Collagen Paste - 6 Month Post-op | Permacol Collagen Paste - 12 Month Post-op
Number analyzed (Participants) | 85 | 76 | 70
units on a scale | -1.0 (3.75) | -1.1 (3.58) | -0.9 (3.75)

5. Secondary Outcome: Patient Satisfaction Between the First and Last Post-operative Visit
Description: Patient satisfaction questionnaire included questions regarding fecal continence and overall satisfaction with the operation.
Time Frame: Between the first and last visits
Population: Number of participants completed a satisfaction questionnaire at least twice.
Measure: Count of Participants; unit: Participants
Arm/Group | First Visit | Last Visit
Number analyzed (Participants) | 85 | 85
Participants
  Very Satisfied | 37 | 44
  Satisfied | 39 | 18
  Dissatisfied | 8 | 18
  Very Dissatisfied | 1 | 5

6. Secondary Outcome: Pain
Description: Pain by VAS (Visual Analog Scale) VAS is a 10-point scale with 0 being no pain and 10 being the most pain.
Time Frame: Baseline, 1 month, 3 months, 6 months and 12 months
Population: Participants include number of patients who completed questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Permacol Collagen Paste - 1 Month Post-op | Permacol Collagen Paste - 3 Month Post-op | Permacol Collagen Paste - 6 Month Post-op | Permacol Collagen Paste - 12 Month Post-op
Number analyzed (Participants) | 98 | 98 | 88 | 79 | 74
Participants
  No Pain (0) | 29 | 45 | 47 | 47 | 53
  Mild Pain (1-3) | 44 | 41 | 33 | 26 | 13
  Moderate Pain (4-6) | 17 | 11 | 7 | 4 | 5
  Severe Pain (7-10) | 8 | 1 | 1 | 2 | 3

ADVERSE EVENTS:
Arm/Group | Permacol Collagen Paste
Serious Adverse Events (participants affected / at risk) | 6/100
Other Adverse Events (participants affected / at risk) | 29/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permacol Collagen Paste (N=100)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal Abscess (Infections and infestations) | 2
Complex regional pain syndrome (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Permacol Collagen Paste (N=100)
Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Anal Fistula (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 6
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Anal abscess (Infections and infestations) | 4
Anal fistula infection (Infections and infestations) | 2
Infected fistula (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
pneumonia (Infections and infestations) | 1
postoperative wound infection (Infections and infestations) | 3
purulent discharge (Infections and infestations) | 1
facial bones fracture (Injury, poisoning and procedural complications) | 1
procedural pain (Injury, poisoning and procedural complications) | 3
Seroma (Injury, poisoning and procedural complications) | 2
Complex regional pain syndrome (Nervous system disorders) | 1
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
breast mass (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
eczema (Skin and subcutaneous tissue disorders) | 1
hypertrophic scar (Skin and subcutaneous tissue disorders) | 1
haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No